CLINICAL TRIAL: NCT06498817
Title: Testing a Scalable Model of the Cholera Hospital-Based Intervention for 7 Days (CHoBI7)
Acronym: CHoBI7
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Research Training and Management International (RTMI) (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); GiveWell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00015070
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Diarrhea Infectious; Cholera
Keywords: randomized controlled trial; Bangladesh; cholera; diarrheal diseases; water, sanitation, and hygiene; healthcare facilities; mobile health; child health
MeSH Terms: conditions — Dysentery; Cholera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Recommendation (Active Comparator): Standard recommendation given by government of Bangladesh on the use of oral rehydration solution (ORS) and a flyer on water treatment and handwashing with soap given at the health facility during the time of diarrhea patient treatment.
  Interventions: Behavioral: Standard Recommendation
- CHoBI7 Scale-Up Program (Experimental): Health promoter delivery of handwashing with soap, water treatment, and safe water storage module in the health facility to diarrhea patients and the patient's household members during the time of treatment. This module includes video testimonials from diarrhea patient households on how the patient benefits from adhering to the promoted behaviors, and a demonstration on how to construct homemade handwashing washing stations. This in-person module is reinforced by weekly voice, interactive voice response, and text messages for three months sent to the mobile phones of diarrhea patient household members from a doctor at diarrhea ward at local hospital.
  Interventions: Behavioral: Standard Recommendation; Behavioral: CHoBI7 Scale-Up Program

INTERVENTIONS:
Behavioral: Standard Recommendation — Standard recommendation given by government of Bangladesh on the use of oral rehydration solution (ORS) and a flyer on water treatment and handwashing with soap given at the health facility during the time of diarrhea patient treatment.
Behavioral: CHoBI7 Scale-Up Program — Health promoter delivery of handwashing with soap, water treatment, and safe water storage module in the health facility to diarrhea patients and the patient's household members during the time of treatment. This module includes video testimonials from diarrhea patient households on how the patient benefits from adhering to the promoted behaviors, and a demonstration on how to construct homemade handwashing washing stations. This in-person module is reinforced by weekly voice, interactive voice response, and text messages for three months sent to the mobile phones of diarrhea patient household members from a doctor at diarrhea ward at local hospital.
  Arms: CHoBI7 Scale-Up Program

SUMMARY:
The findings from previous recent randomized controlled trials of The Cholera Hospital Based Intervention for 7 Days (CHoBI7) demonstrated that this intervention was effective in significantly reducing symptomatic cholera infections, diarrheal disease, and stunting among young children in intervention households, and had significant sustained impacts on handwashing with soap behaviors and improved water quality 12 months post intervention. Therefore, the investigators next step in the transition to scale is to: (1) To tailor the CHoBI7 program for delivery in rural health facilities and market test the CHoBI7 Program to determine the feasibility of providing a modified water, sanitation, and hygiene (WASH) package with only a soapy water bottle and chlorine tablets in both urban and rural settings through formative research and engagement of key stakeholders (Formative Research Phase); and (2) To evaluate the effectiveness of delivering the CHoBI7 program in district hospitals and sub-district health complexes in rural areas in terms of increases in WASH behaviors and decreases in diarrheal disease by conducting a randomized controlled trial (RCT) (Intervention Implementation and Evaluation Phase).

DETAILED DESCRIPTION:
Diarrhea is the second leading cause of death in children under 5 years of age globally, causing an estimated 800,000 deaths annually. Previous studies have identified lack of caregiver hand washing with soap and treatment of household drinking water, poor water storage practices, and lack of caregiver knowledge of diarrhea prevention as important risk factors for diarrheal disease in pediatric populations. Water, sanitation, and hygiene (WASH) interventions promoting household chlorination of drinking water and hand washing with soap have the potential to reduce diarrheal disease incidence in children less than five years of age an estimated 30 to 40%. However, there has been limited success in encouraging households to sustain these behaviors over time. Furthermore, community-based WASH interventions are expensive and often difficult to implement in an urban context in low resource settings.

Previous studies have found that at the time of a severe illness such as cholera outbreaks, households have higher perceived severity and benefits of water treatment. In Madagascar an intervention which promoted the use of chlorine and 20 liter jerry cans reached peak sales during the high season for cholera. Consistent findings were observed in Zambia where sales of a water treatment product called Clorin significantly increased during a cholera epidemic. Furthermore in Dhaka, Bangladesh, the use of a community level point of use chlorine dispenser peaked after cholera deaths in a slum area of the city. Therefore admission at a health care facility for the treatment of severe diarrhea could potentially serve as an ideal opportunity to promote WASH interventions on improved water treatment and hygiene practices

The research team developed a Hospital Based WASH intervention which is entitled CHoBI7 (Cholera Hospital-Based Intervention for 7 days). Chobi means "picture" in Bangla for the pictorial WASH module delivered as part of the program. The CHoBI7 intervention was initially designed to reduce cholera infection among family members of hospitalized cholera cases during the one week high risk period after the case presents at the hospital. This Hospital Based WASH intervention is disseminated by health facility based promoters to hospitalized diarrhea patients and the family members and includes: (1) A pictorial module on diarrhea transmission and prevention, and (2) A diarrhea prevention package which contains chlorine tablets for water treatment, a soapy water bottle and a hand washing station, and a sealed water vessel to ensure safe water storage. The findings from previous recent randomized controlled trials of The Cholera Hospital Based Intervention for 7 Days (CHoBI7) demonstrated that this intervention was effective in significantly reducing symptomatic cholera infections, and had significant sustained impacts on hand washing with soap behaviors and improved water quality 12 months post intervention.

In an effort to build evidence to take the CHoBI7 intervention to scale in Bangladesh, the investigators partnered with the Bangladesh Ministry of Health and Family Welfare (MoHFW) to develop and evaluate scalable approaches for CHoBI7 intervention delivery. The CHoBI7 intervention was broaden during this time to include diarrhea patients of all etiology not just cholera. In addition, the investigators developed the CHoBI7 WASH mobile health (mHealth) program, to serve as a low cost scalable approach to reinforce the CHoBI7 WASH pictorial module delivered in the health facility without the need for home visits. After health facility delivery of the CHoBI7 pictorial module by a health worker, diarrhea patient households receive weekly voice and text messages from the CHoBI7 mHealth program over a 12 month period. The CHoBI7 WASH mHealth program significantly decreased diarrhea and stunting among young children, and lead to sustained handwashing with soap practices and improved stored drinking water quality during the 12 month surveillance period in an urban setting in Dhaka, Bangladesh during the investigators recent randomized controlled trial.

The investigators goal for this study is to develop a scalable version of the CHoBI7 program that can be delivered in district hospitals and sub-district health complexes in rural and urban Bangladesh. This scalable version of the CHoBI7 program will provide only a soapy water bottle and chlorine tablets, and encourage households to construct a handwashing station themselves using items in the homes

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea patients presenting with three or more loose stools over a 24h period
* Having no running water inside of the patient's home
* Plan to reside in current residence for the next 3 months
* Have a child <5 years in the patient's household
* Have a working mobile phone in the household

Exclusion Criteria:

* No one will be excluded because of age, sex, religion, or sexual preference

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Handwashing with soap at stool and food related events | 3 months
  Rate of patient household members handwashing with soap at stool and food related events measured measured using a 5 hour structured observation tool in the household using form developed by the investigators.
Number of constructed homemade handwashing stations | 3 months
  Household construction of homemade handwashing station

SECONDARY OUTCOMES:
Number of participants with diarrhea | 3 months
  Number of participants with self-reported or caregiver reported diarrhea (3 or more loose stools for a 24 hour period)
Amount of free chlorine concentration in stored drinking water | 3 months
  mg/Liter
Number of stored drinking water samples with E. coli | 3 months
  Number of stored drinking water samples with E. coli
Water, sanitation, and hygiene (WASH) psychosocial factors | 3 months
  Water, Sanitation, and Hygiene (WASH) psychosocial risk factor questionnaire. 5-point scale (0 = [almost] never/0-1 times out of 10-1 = [almost] always/9-10 times out of 10). with higher scores indicating higher handwashing frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Marie George, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Manikganjg Sadar (District) Hospital, Mānikganj, Bangladesh

IPD SHARING:
Plan to Share IPD: No